CLINICAL TRIAL: NCT02357407
Title: Development of an Adjustment Assistance Tool Dosage of Fluoroquinolones in a Population Pharmacokinetic Model
Acronym: FLUO-POP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-004193-4; 35RC14_9179 (Other: CHU Rennes)
Record Dates: First submitted 2015-01-16; First posted 2015-02-06 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Infection
Keywords: fluoroquinolones; pharmacokinetic; infections
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection; Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients in intensive care (Experimental): 30 patients in intensive care treated with ciprofloxacin IV
  Interventions: Drug: Patients in intensive care : infection treated with ciprofloxacin IV
- Osteoarticular infected patients (Experimental): 30 patients in orthopedics treated with oral ofloxacin
  Interventions: Drug: Osteoarticular infected patients : infection treated with oral ofloxacin

INTERVENTIONS:
Drug: Patients in intensive care : infection treated with ciprofloxacin IV — 8-10 samples per patients on day-4 of their treatment
  Other Names: Blood samples
  Arms: Patients in intensive care
Drug: Osteoarticular infected patients : infection treated with oral ofloxacin — 8-10 samples per patients on day-4 of their treatment
  Other Names: Blood samples
  Arms: Osteoarticular infected patients

SUMMARY:
Fluoroquinolones (FQ) are among pivotal antibiotic treatments in difficult-to-treat infections. Their efficacy has been shown to be linked to the ratio area under the curve (AUC) of their plasma concentrations over the minimum inhibitory concentration (MIC) of the bacteria treated. Eventually, Forrest et al., reported in gram-negative infections that an AUC/MIC above 125 conducted to a 80 to 90% clinical success whereas success decrease to 30 to 40% in patients with an AUC/MIC below this threshold. These results have been reproduced recently by Zelenitsky et al. in intensive care unit (ICU) patients with threshold similar to the one obtained by Forrest et al. Lastly, elevated concentrations of FQ should be related with the onset of adverse events. Thus, therapeutic drug monitoring (TDM) of FQ appears of potential interest, particularly in case of severe infections (intensive care unit (ICU) patients) or complicated and cost-related infections (osteoarticular infected (OAI) patients), with an increasing level of evidence of its use.

However, FQ TDM requires access to the full AUC of the drug with the need of many samples drawn to patients. This appears to be irreconcilable with clinical practice but can be achieved using population pharmacokinetic (PkPop) modelling. PkPop allows estimating pharmacokinetic parameters of the drug by introducing covariates (demographic, biological, clinical…) and modelling inter-individual pharmacokinetic variability. The model created allows then accessing to individual parameters of patients and thus, estimating concentrations and AUC of the FQ. This approach may also be used in clinical practice to determine a limited sampling strategy allowing an adequate estimation of AUC with a minimum of samples.

DETAILED DESCRIPTION:
Open, prospective, monocentric pharmacokinetic study

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients in intensive care : Infection treated with ciprofloxacin IV
* Osteoarticular infected patients : infection treated with oral ofloxacin
* Written consent to participate in the study

Exclusion Criteria:

* Pregnancy
* Adults subject to legal protection or deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration measurement of ciprofloxacin and ofloxacin | on day-4 of their treatment (steady-state)
  measurement between 2 administrations (8-10 samples per patients)

SECONDARY OUTCOMES:
Demographic data | on day-4 of their treatment (steady-state)
Biological data | on day-4 of their treatment (steady-state)
Clinical data | on day-4 of their treatment (steady-state)
AUC | on day-4 of their treatment (steady-state)
MIC | on day-4 of their treatment (steady-state)
Cmax | on day-4 of their treatment (steady-state)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BL Laviolle, MD/PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Result] Lemaitre F, Fily F, Foulquier JB, Revest M, Jullien V, Petitcollin A, Tattevin P, Tron C, Polard JL, Verdier MC, Comets E, Huten D, Arvieux C, Bellissant E, Laviolle B. Development of a dosing-adjustment tool for fluoroquinolones in osteoarticular infections: The Fluo-pop study. Biomed Pharmacother. 2021 Oct;142:112053. doi: 10.1016/j.biopha.2021.112053. Epub 2021 Aug 19. PMID 34435591